CLINICAL TRIAL: NCT01464086
Title: LIFSCREEN : Evaluation of Whole Body MRI for Early Detection of Cancers in Subjects With P53 Mutation (Li-Fraumeni Syndrome)
Acronym: LIFSCREEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CSET2011/1748
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Li Fraumeni Syndrome
Keywords: patients with Li Fraumeni syndrome
MeSH Terms: conditions — Li-Fraumeni Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard arm (No Intervention): standard follow-up
- Intensive follow-up (Experimental): Standard follow-up plus whole body MRI at inclusion, one and two years
  Interventions: Other: whole body MRI

INTERVENTIONS:
Other: whole body MRI — whole body MRI at inclusion, one and two years
  Arms: Intensive follow-up

SUMMARY:
The purpose of this study is to compare the diagnostic efficacy of two follow-up schedules for the early detection of cancers in the population under study on cancer incidence at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* P53 mutation

Ages: 5 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-10-27 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
cancer incidence | 3 years
  cancer incidence during the first 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Caron O, Frebourg T, Benusiglio PR, Foulon S, Brugieres L. Lung Adenocarcinoma as Part of the Li-Fraumeni Syndrome Spectrum: Preliminary Data of the LIFSCREEN Randomized Clinical Trial. JAMA Oncol. 2017 Dec 1;3(12):1736-1737. doi: 10.1001/jamaoncol.2017.1358. PMID 28772306